CLINICAL TRIAL: NCT01528163
Title: Randomized Phase II Study of Cabazitaxel Versus Methotrexate in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck Previously Treated With Platinum-based Therapy.
Brief Title: Study Comparing Two Treatments in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Acronym: RACATREX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 2011-01; 2011-001938-42 (EudraCT Number)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and neck; Squamous cell carcinoma; Randomized; palliative treatment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — cabazitaxel; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabazitaxel (Experimental): Cabazitaxel (XRP6258) is a new taxoid, which promotes tubulin assembly in vitro and stabilizes microtubules against cold-induced depolymerization as efficiently as docetaxel
  Interventions: Drug: Cabazitaxel
- Methotrexate (Active Comparator): Methotrexate is the historical control and has been widely used in SCCHN for palliation.
  This medication is an antimetabolite and antifolate drug. It acts by inhibiting the metabolism of folic acid.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Cabazitaxel — from 20 mg/m2 to 25 mg/m2. Intravenous injection every three weeks.
  Other Names: Jevtana
  Arms: Cabazitaxel
Drug: Methotrexate — From 40 mg/m2 (first cycle) to 50 mg/m2. Intravenous injections every three weeks.
  Other Names: Emthexate
  Arms: Methotrexate

SUMMARY:
In this clinical trial, the investigators want to know if cabazitaxel is more effective than methotrexate for patients with recurrent or metastatic squamous cell carcinoma of the head and neck in palliative treatment.

DETAILED DESCRIPTION:
The principal aim is to evaluate the efficacy of cabazitaxel in patients with palliative head and neck previously treated with platinum-based therapy.

The study design is a non comparative randomized phase II trial: ARM 1: cabazitaxel (20 mg/m2, every 3 weeks) versus ARM 2 methotrexate (40 mg/m2, weekly). Cabazitaxel dose will be increased to 25mg/m2 for the second and subsequent cycles, in the absence of non-hematological AE > grade 2 and hematological AE > grade 3 during the first cycle. (maximum 10 cycles). The aim of the randomization is to offer a valid internal control group by avoiding possible selection bias. However, results obtained in the two treatment group will not be formally compared as this is not the objective of a phase II study.

Tumor check-up will be performed every 9 weeks. Treatment will be continued until disease progression or unacceptable toxicities according to the patient or the investigator. A maximum of 10 cycles of cabazitaxel will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent and/or metastatic head and neck squamous cell carcinoma not amenable to curative treatment with surgery and/or chemotherapy and/or radiation.
2. At least one measurable lesion by MRI or CT-scan according to RECIST 1.1.
3. Progressive disease within 1 year after first line platinum-based chemotherapy given either as a part of the multimodal curative treatment or in the palliative setting.
4. ECOG performance status 0 -2, in stable medical condition
5. Patients must have an expected survival of at least 3 months
6. Paraffin-embedded tumor tissue available for immunohistochemistry but not mandatory
7. Patients must be over 18 years old and must be able to give written informed consent.
8. Women of child-bearing age or sexually active female patients with reproductive potential must have a negative pregnancy test (serum or urine within the 7 days prior to enrollment).
9. Patients must have adequate organ function (Hemoglobin ≥ 9 g/100 ml, Neutrophils ≥ 1,500/mm3, Platelets ≥ 100,000/mm3, total bilirubin <1 time the upper limit of normal (ULN) for age, serum alanine aminotransferase (ALT) < 1.5 1.5 x ULN for age, aspartate aminotransferase (AST) < 1.5 ´ ULN for age , serum creatinine <1.5 x ULN for age.
10. Signed informed consent prior to beginning protocol specific procedure.
11. Sexually active patients must use effective contraception during the period of therapy and up to 150 days after the last treatment dose. Acceptable contraception includes, but is not limited to: oral hormone therapy, partner vasectomy, or double barrier contraception (which is defined as a male condom plus spermicide in combination with either a female condom, or diaphragm, or cervical cap or intrauterine device)

Exclusion Criteria:

1. Non-squamous head and neck cancer
2. Nasopharynx cancer
3. More than two lines of chemotherapy for palliative treatment
4. Surgery or investigational drugs or chemotherapy within 4 weeks before study inclusion. Curative radiation therapy (60-70 Gy) within 8 weeks. For palliative radiation therapy (i.e 8 Gy on a painful lesion) no delay is needed.
5. Previous treatment with cabazitaxel
6. Significant active cardiac disease including: uncontrolled high blood pressure according to the CTCAE 4 grading, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, or serious cardiac arrhythmias
7. Other uncontrolled illnesses (active infections requiring antibiotics, bleeding disorders, uncontrolled diabetes …)
8. Previous malignancy from which the patient has been disease-free for < 5years, as other than SCCHN.
9. Previous treatments with taxanes and/or anti-EGFR therapy are not an exclusion criteria.
10. Active grade > 2 peripheral neuropathy
11. Active grade > 2 stomatitis
12. Known brain or leptomeningeal involvement
13. History of severe hypersensitivity reaction (> grade 3) to polysorbate 80 containing drugs
14. Concurrent or planned treatment with strong inhibitors of cytochrome P450 3A/5. A one-week washout period is necessary for patients who are already on these treatments.
15. Organic brain syndrome or significant psychiatric abnormality that would preclude participation in the full protocol and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Efficacy | 18 weeks
  Determine the efficacy of cabazitaxel in patients with head and neck cancer in terms of progression-free survival rate at 18 weeks.

SECONDARY OUTCOMES:
Safety profile | 18 weeks
  Determine the safety profile of cabazitaxel in patients with head and neck cancer: adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, PhD, Principal Investigator — Centre du Cancer, Cliniques universitaires Saint-Luc
Locations (16):
- Belgium (15):
  - Clinique Saint-Pierre, Ottignies, Brabant Wallon
  - Cliniques universitaires Saint-Luc, Centre du Cancer, Oncologie Médicale, Brussels, Brussels Capital
  - RHMS Baudour, Baudour, Hainaut
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Hôpital de Jolimont, Haine-Saint-Paul, Hainaut
  - CHU Tivoli Centre René Goffin, La Louvière, Hainaut
  - CHU Ambroise PARE, Mons, Hainaut
  - CHU de Charleroi site Vésale, Montigny-le-Tilleul, Hainaut
  - Centre Hospitalier Wallonie Picarde, Tournai, Hainaut
  - CHU de Mont Godinne, Yvoir, Namur
  - Universitair Ziekenhuis Brussel (Campus Jette), Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - CHR Citadelle, Liège
  - CHU de Liège Sart Tilman, Liège
  - Clinique et Maternité Sainte-Elisabeth, Namur
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Machiels JP, Van Maanen A, Vandenbulcke JM, Filleul B, Seront E, Henry S, D'Hondt L, Lonchay C, Holbrechts S, Boegner P, Brohee D, Dequanter D, Louviaux I, Sautois B, Whenham N, Berchem G, Vanderschueren B, Fontaine C, Schmitz S, Gillain A, Schoonjans J, Rottey S. Randomized Phase II Study of Cabazitaxel Versus Methotrexate in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck Previously Treated With Platinum-Based Therapy. Oncologist. 2016 Dec;21(12):1416-e17. doi: 10.1634/theoncologist.2016-0296. Epub 2016 Nov 30. PMID 27903924